CLINICAL TRIAL: NCT07234630
Title: Role of Fibrinolytic Activity in Neoplastic Pathologies Complicated by Coagulopathy
Acronym: NEO-COAG
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9558
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Neoplasms; Solid Tumor Metastatic Cancer Advanced Cancer; Disseminated Intravascular Coagulation
MeSH Terms: conditions — Hematologic Neoplasms; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Hematological malignancies with large tumor masses: * Acute myeloblastic or lymphoblastic leukemia with leukocyte count (or blasts) >50G/L in peripheral blood, or
  * Lymphoma documented by tissue biopsy, with biological tumor lysis syndrome, diagnosed according to Cairo and Bishop criteria.
  Interventions: Biological: An additional volume of blood will be drawn as part of routine follow-up care
- Group 2: Locally advanced or metastatic solid tumors with DIC: * Prostatic adenocarcinoma
  * Malignant pancreatic or biliary tract tumor (cholangiocarcinoma),
  * Scheduled complex hepatobiliary carcinological surgery,
  * Metastatic adenocarcinoma of the digestive tract.
  Interventions: Biological: An additional volume of blood will be drawn as part of routine follow-up care
- Group 3: Control group (free of neoplastic pathology, with well-studied coagulopathy): Defined according to Sepsis-criteria
  Interventions: Biological: An additional volume of blood will be drawn as part of routine follow-up care

INTERVENTIONS:
Biological: An additional volume of blood will be drawn as part of routine follow-up care — The biological samples collected correspond to blood samples taken from venous or arterial catheters inserted at the time of admission as part of routine care. The total volume of blood collected at D1 and D7 was 18.5 mL (3 x 4 mL citrate tubes, 1 x 4 mL EDTA tube and 1 x 2.5 mL Paxgene tube). The volume of blood drawn at D3 was 16 mL (3 x 4 mL citrated tubes, one 4 mL EDTA tube).
  Samples are immediately analyzed in the hematology/hemostasis laboratory for NETs and hemostasis, with the remaining portion of the tube centrifuged before plasma is frozen at -80°C for plasma analysis. The Paxgene tube can be used for non-identifying genetic analyses.

SUMMARY:
The aim of this research is to measure fibrinolytic activity in neoplastic pathologies in order to provide preliminary data on which to base a future, larger-scale study to determine predictive markers of complication in order to improve patient management.

Primary purpose: measure plasminogen concentration on day 1 in subjects diagnosed with malignant hematological disease, solid tumors, or septic shock, with coagulopathy.

Secondary purpose:

* Estimate the difference in plasminogen concentration at D1 in patients with coagulopathy between subjects with a diagnosis of haematological malignancy and those with solid tumor
* Estimate the difference in plasminogen concentration at D1 in patients with coagulopathy between subjects with a diagnosis of haematological malignancy and those with septic shock
* Estimate the difference in plasminogen concentration on Day 1 in patients with coagulopathy between subjects with a diagnosis of solid tumor and those with septic shock.

In the 3 groups, subjects with a diagnosis of haematological malignancy, solid tumor, septic shock, presenting with coagulopathy:

* Evaluate the correlation between the concentration of circulating plasminogen active on Day 1 and the occurrence of a bleeding complication within 28 days of admission to critical care.
* Evaluate the correlation between the concentration of circulating plasminogen active on Day 1 and the occurrence of a thrombotic complication, within 28 days of admission to critical care.
* Evaluate the predictive performance of circulating active plasminogen concentration on Day 1 in the need for extra renal purification within 28 days of admission to critical care.
* Estimate the differences at each time point (D1, D3, D7) in haemostasis markers and markers of fibrinolytic activity and its regulation.

Assess the link between fibrinolytic activity and :

* The diagnosis of disseminated intravascular coagulation (DIC),
* The risk of haemorrhage
* Risk of organ failures
* Thrombotic risk
* Risk of organ failure
* Neutrophile activation and circulating NETs levels

ELIGIBILITY:
Inclusion Criteria:

For all groups:

* Age > 18 years
* Patient hospitalized in Emergency Medicine, Intensive Care Medicine or Hematology/Oncology Intensive Care, Hematology/Oncology Service or Hepatobiliary and Digestive Surgery Service
* Coagulopathy defined by the combination of thrombocytopenia (< 100 G/L) and increased INR (>1.2)

Group 1: Malignant hemopathies with large tumor masses:

* Acute myeloblastic or lymphoblastic leukemia with leukocyte count (or blasts) >50G/L in peripheral blood, or
* Lymphoma documented by tissue biopsy, with biological tumor lysis syndrome, diagnosed according to Cairo and Bishop criteria (3).

Group 2: Locally advanced or metastatic solid tumors with DIC:

* Prostatic adenocarcinoma
* Malignant pancreatic or biliary tract tumor (cholangiocarcinoma),
* Scheduled complex hepatobiliary carcinological surgery,
* Metastatic adenocarcinoma of the digestive tract.

Group 3: Control group (free of neoplastic pathology, with well-studied coagulopathy): Septic shock

Exclusion Criteria:

* Patient under protective supervision (guardianship or curatorship)
* Pregnant women
* Patients weighing less than 50 kg
* Patient already included in the study
* Congenital hemostasis disorders
* Active bleeding at the time of inclusion
* Patient with cirrhosis
* Patients receiving curative anticoagulation therapy
* Patients with a spontaneous INR > 1.2 in a previous blood test in a context of fibrinolytic insufficiency
* Each group is exclusive of the other, for example :

For Group 1 (Neoplastic pathologies): Presence of documented sepsis at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The populations studied are neoplasia carriers with coagulopathy defined by the association of thrombocytopenia (<100G/L) and increased INR (>1.2).
  Adult patients hospitalized in Emergency Medicine, Intensive Care Medicine or Hepatobiliary and Digestive Surgery Service.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Plasminogen measurement at D1 in hematologic malignancy, solid tumor and septic shock groups. | Day 1
  The biological samples collected correspond to blood samples taken from venous or arterial catheters inserted at the time of admission as part of routine care.

SECONDARY OUTCOMES:
Measurement of various haemostasis markers | Day 1, 3 and 7
  Measurement of platelet count, PT/INR, aPTT, fibrinogen, factor V, D-dimers, antithrombin III, factor VIII
Measurement of markers of fibrinolytic activity and its regulation | Day 1, 3 and 7
  Assay of t-PA, u-PA, PAI-1, u-PAR, plasmin activity
Analysis of parameters closely associated with serum NET assays | Day 1, 3 and 7
  Measurement of neutrophil fluorescence, circulating nucleosomes

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Clere-Jehl, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No